CLINICAL TRIAL: NCT00288210
Title: Randomized Study Of Sirolimus Eluting Stent Vs Conventional Stent In Acute Myocardial Infarction Acronym SESAMI
Brief Title: Sirolimus Eluting Stenting in Acute Myocardial Infarction
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: San Camillo Hospital, Rome (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 183/2003
Record Dates: First submitted 2006-02-06; First posted 2006-02-07 (Estimated); Last update posted 2006-02-10 (Estimated); Status verified 2006-02

CONDITIONS: Myocardial Infarction
Keywords: Myocardial Infarction; Stents; Sirolimus; abciximab
MeSH Terms: conditions — Myocardial Infarction

INTERVENTIONS:
Procedure: Primary angioplasty in acute myocardial infarction

SUMMARY:
The incidence of stent restenosis in the setting of primary angioplasty is particularly high, reaching a rate of 27% In the last years the introduction of drug-eluting stents has drastically reduced the incidence of restenosis in patients not requiring urgent revascularization. Whether drug-eluting stenting might constitute the new optimal therapy for patients with an acute myocardial infarction is unknown. To be able to answer this question, we designed a randomized trial in which patients with an acute myocardial infarction eligible for treatment with primary angioplasty and abciximab were randomized to receive either a rapamicine-eluting stent or a conventional bare stent.

DETAILED DESCRIPTION:
The treatment of acute myocardial infarction has evolved dramatically in the last decade. Coronary angioplasty with stent implantation in conjunction with an optimal antitrombotic therapy as abciximab is now considered current standard therapy However, the incidence of stent restenosis in the setting of primary angioplasty remains particularly high, reaching a rate of 27%. A high restenosis rate causes a high re-hospitalization rate for target vessel revascularization and an ensuing increase in cost.In the last years the introduction of drug-eluting stents has drastically reduced the incidence of restenosis in patients not requiring urgent revascularization. This reduced incidence of restenosis occurs without an increase in adverse clinical events over conventional stents and has a very low rate of stent subacute thrombosis. Whether this combination of drug-eluting stents and abciximab might constitute the new optimal therapy for patients with an acute myocardial infarction is unknown. To be able to answer this question, we designed a one year coronary angiographic study in which patients with an acute myocardial infarction eligible for treatment with primary angioplasty and abciximab were randomized to receive either a rapamicine-eluting stent or a conventional bare stent.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria were an age of more than 18 years, the presence for at least 30 minutes but less than 12 hours of symptoms consistent with acute myocardial infarction, and the presence of ST-segment elevation in at least two contiguous leads or left bundle-branch block.

-

Exclusion Criteria:

Patients were excluded if they were in cardiogenic shock (defined as systolic blood pressure of less than 80 mm Hg for more than 30 minutes or the need for intravenous pressors or intraaortic-balloon counterpulsation); had a history of bleeding diathesis; had a history of leukopenia, thrombocytopenia, or severe hepatic or renal dysfunction; had a noncardiac illness associated with a life expectancy of less than one year; were participating in another study; or were unable to give informed consent owing to prolonged cardiopulmonary resuscitation.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-03; Study Completion 2006-03

PRIMARY OUTCOMES:
The primary end point for the trial was the binary restonis at one year angiographic follow-up

SECONDARY OUTCOMES:
Secondary end points included a composite of
MACE including death, Q-wave and non-Q-wave infarction, emergent bypass surgery, or repeat TLR at 30 days and 12 months after the index procedure

CONTACTS AND LOCATIONS:
Overall Officials: Roberto Violini, MD, Study Chair — Cardiologia Interventistica Ospedale San Camillo Roma; Maurizio Menichelli, MD, Principal Investigator — Cardiologia Interventistica Ospedale San Camillo Roma
Locations (1):
- Cardiologia Interventistica Ospedale San Camillo, Roma, Roma, Italy

REFERENCES:
- [Derived] Menichelli M, Parma A, Pucci E, Fiorilli R, De Felice F, Nazzaro M, Giulivi A, Alborino D, Azzellino A, Violini R. Randomized trial of Sirolimus-Eluting Stent Versus Bare-Metal Stent in Acute Myocardial Infarction (SESAMI). J Am Coll Cardiol. 2007 May 15;49(19):1924-30. doi: 10.1016/j.jacc.2007.01.081. Epub 2007 Apr 30. PMID 17498576